CLINICAL TRIAL: NCT01110954
Title: Evaluation of the Suitability of PD L 506 for Intraoperative Visualisation of Palpable and Nonpalpable Breast Cancer Tissue
Brief Title: Fluorescence-guided Resection in Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: photonamic GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MK01
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Breast Tumour
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PD L 506 2nd dose (Active Comparator): Different dosage
  Interventions: Drug: PD L 506
- PD L 506 (Experimental)
  Interventions: Drug: PD L 506

INTERVENTIONS:
Drug: PD L 506 — Two different doses will be compared

SUMMARY:
This is an explorative phase II study to investigate the suitability of PD L 506 in the specific intra-operative detection of breast tumour tissue.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Caucasian female postmenopausal patients
* Patients with histologically confirmed primary palpable and nonpalpable breast cancer sized up to 5 cm (T1 - T2)

Exclusion Criteria:

* Suspicious lymphogenic metastases (cN1-3)
* Acute or chronic hepatic diseases
* Manifest renal diseases with renal dysfunction
* Relevant cardiac disease
* Preceding therapy of breast tumour under investigation
* Patients with multiple attempts of hook-wire placement in preparation of surgery
* Dementia or psychic condition that might interfere with the ability to understand the study and thus give a written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2012-07-19 (Actual); Study Completion 2012-12-20 (Actual)

PRIMARY OUTCOMES:
Fluorescence intensity in breast cancer tissue | 3 h after intake of study medication

SECONDARY OUTCOMES:
Laboratory data and adverse events | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Munich, Germany